CLINICAL TRIAL: NCT06619093
Title: Relationship Between Biological Phenotype, Clinical Severity of Sickle Cell Disease, and Blood Coagulation
Acronym: DREPA COAG
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (UCBL1) UR7424 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0679
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Hemolysis; Coagulation; Red blood cell; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hemolysis; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High hemolytic group: Lactate Dehydrogenase Level > 484 IU/L
  Interventions: Other: blood sampling
- Low hemolytic group: Lactacte Dehydrogenase Level less or equal to 484 IU/L
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — 3 additional citrate tubes (2.7mL)

SUMMARY:
Sickle cell disease is characterized by chronic hemolytic anemia and blood rheological alterations. In addition, blood coagulation abnormalities have been reported in patients with sickle cell disease and hemolysis-derived products could be involved. The investigators hypothesized that patients with sickle cell disease and severe hemolysis (Lactate Dehydrogenase level > 484 IU/L) could have an increased risk of hypercoagulable state and subsequent thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8 years or older
* Under clinical follow-up for a diagnosis of sickle cell disease, specifically genotypes S/S, S/beta0, or S/C
* Patient covered by a social security or equivalent health insurance plan
* Collection of the non-opposition for adults
* Information of the minor and collection of the non-opposition from both parents

Exclusion Criteria:

* Patient who has undergone a transfusion or therapeutic phlebotomy within the 3 months prior to inclusion
* Patient participating in another interventional research protocol that may interfere with the present protocol (at the investigator's discretion)
* Patient under guardianship, curatorship, or legal protection
* Patient subject to a legal protection measure
* Person admitted to a health or social care institution for purposes other than research

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sickle cell disease, followed regularly by the Sickle Cell Center of Lyon Hospitals (Hospices Civils de Lyon).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall coagulation activity | Baseline
  To compare the overall coagulation activity (measurement of in vitro clot formation by rotary thromboelastometry (ROTEM)) between sickle cell patients with a severe haemolytic phenotype and those with a less severe haemolytic phenotype.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Insitut Hématologique et Oncologique Pédiatrique (IHOPe), Lyon
  - Service de Médecine Interne - Hôpital Edouard Herriot, Lyon

IPD SHARING:
Plan to Share IPD: Undecided